CLINICAL TRIAL: NCT01325961
Title: Medico-economic Evaluation Comparing Conformal Radiotherapy With Intensity Modulation (IMRT) Performed by, Helical Tomotherapy (Hi Art) and Dynamic Arc Therapy (RapidArc, VMAT) in Cancers With Pelvic Lymph Node Irradiation (Prostate, Cervix, Anal Canal)
Brief Title: Medico-economic Evaluation Comparing Intensity-Modulated Radiation Therapy (IMRT) Performed by Helical Tomotherapy and Dynamic Arc Therapy in Prostate, Cervical and Anal Canal Cancers
Acronym: RCMI PELVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BRD 10/12-O
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2016-08

CONDITIONS: Prostate Cancer; Cervical Cancer; Anal Canal Cancers
Keywords: prostate, cervical and anal canal cancers with pelvic lymph node irradiation
MeSH Terms: conditions — Prostatic Neoplasms; Uterine Cervical Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy

SUMMARY:
The aim of the study is a medico-economic evaluation to estimate a cost differential between three modalities of Intensity-Modulated Radiation Therapy for cancers of the prostate, cervix and anal canal with pelvic lymph node irradiation : treatment with helical Tomotherapy and dynamic arc therapy using two different technologies: RapidArc or VMAT.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance index ≤ 2
* Age > 18 years
* histologically proven carcinoma: Anal canal cancer locally advanced (> 4 cm and / or N1 to N3) under irradiation on pelvic and inguinal lymph nodes with concurrent chemotherapy. The boost with brachytherapy are accepted Prostate cancer with pelvic lymph nodes and radiation or hormone therapy Cervical Cancer under a purely medical treatment involving irradiation on pelvic lymph nodes and primary tumor with concurrent chemotherapy without surgery. The Boost by external radiotherapy or brachytherapy are accepted.
* The investigator must ensure that the patient has not expressed its opposition to participate in this study. The signing of a consent form is optional;

Exclusion Criteria:

* History of invasive cancer other than basal cell carcinomas.
* Indication of re-irradiation
* para-aortic radiotherapy associated with pelvic irradiation.
* post-operative radiotherapy.
* geographical distance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Medico-economic study : medical cost differential between 3 ways of Radiotherapy by IMRT (helical tomotherapy and dynamic arc therapy : RapidArc and VMAT). | 2 months
  Costs of the devices, maintenance costs ; personnel costs directly related to the medical therapeutic procedure (physicians, medical physicists, dosimetry, technicians).

SECONDARY OUTCOMES:
Others economic criteria | 2 months
  * the estimation of the cost differential by individualizing the preparation phase and phase radiation
  * the analysis of the possible impact of learning in helical tomotherapy and dynamic arc therapy with VMAT and RapidArc measured on direct costs (depending on the age of implantation and equipment)
clinical response and safety of the treatment by radiotherapy | 18 Months (cervix and canal anal) or 36 months (prostate)
  * Assess the skin and mucosal toxicity (acute, delayed) : CTCAEv3
  * Assess the prognostic factors of onset of toxicity
  * Assess oncological results

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Assistance publique des Hôpitaux de Marseille, Marseille
  - Hôpital Clinique Claude Bernard, Metz
  - Groupe Oncorad, Montauban
  - Centre Val d'Aurelle, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Institut Curie, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Groupe Oncorad, Toulouse